CLINICAL TRIAL: NCT06630468
Title: The Effect of Task-oriented Occupational Therapy Intervention on Occupational Performance, Occupational Balance and Quality of Life Among Individuals with Chronic Stroke
Brief Title: Task-Oriented Occupational Therapy Approach in Chronic Stroke: Performance, Balance, Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Zeynep Şule Erkuvan, Occupational Therapist, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOOT_OT_STROKE; Kayseri city hospital (Other: Kayseri city hospital)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2022-12

CONDITIONS: Chronic Stroke; Occupational Therapy; Occupational Balance; Upper Extremity
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator was blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Task-oriented occupational therapy (TOOT) (Experimental): The task-oriented occupational therapy intervention was applied to individuals in the TOOT group in the form of 30-minute sessions, 5 consecutive days a week, over 4 weeks.
  Interventions: Other: Task-oriented occupational therapy (TOOT)
- Control group (Active Comparator): Routine upper-extremity-based occupational therapy intervention was applied to individuals in the TOOT group in the form of 30-minute sessions, 5 consecutive days a week, over 4 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Task-oriented occupational therapy (TOOT) — The task-oriented occupational therapy intervention was applied to individuals in the TOOT group in the form of 30-minute sessions, 5 consecutive days a week, over 4 weeks.
  Other Names: TOOT
  Arms: Task-oriented occupational therapy (TOOT)
Other: Control group — Routine upper-extremity-based occupational therapy intervention was applied to individuals in the TOOT group in the form of 30-minute sessions, 5 consecutive days a week, over 4 weeks.
  Arms: Control group

SUMMARY:
Chronic stroke is a neurological disorder that leads to long-term disability and functional impairments in motor, sensory, cognitive, and speech functions, persisting beyond six months after the stroke incident. The purpose of this study was to investigate the effects of task- oriented occupational therapy intervention on occupational performance, occupational balance, and quality of life in individuals with chronic stroke. The study included 30 individuals with chronic stroke aged between 18 and 65, who were divided into two groups:

the task-oriented occupational therapy intervention group (TOOT) (n=15) and the control group (n=15). The participants in the TOOT group received task-oriented occupational therapy intervention in 30-minute sessions, five days a week, for four weeks, while the control group received routine upper-extremity-based occupational therapy intervention in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old,
* completed the acute phase of stroke
* experienced ischemic and/or hemorrhagic stroke
* had <=21 scores of Montreal Cognitive Assessment (MoCA)
* had <= 15 scores of the Rivermead Motor Assessment (RMA)
* had a motor stage of the hand and upper extremity motor stage level 3 or higher of the Brunnstrom Stages of Motor Recovery
* had scoring 2 or lower on the Modified Ashworth Scale for muscle tone around the shoulder, elbow, and wrist were included into the study.

Exclusion Criteria:

* Had an orthopedic problem affecting the upper extremity
* had undergone surgery in the past 6 months
* had a diagnosis related to a psychotic disorder.

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | From enrollment to the end of treatment at 4 weeks
  The task was used to evaluate occupational performance, developed by the Canadian Association of Occupational Therapists, the Canadian Occupational Performance Measure is used to identify problems in activity performance, measure changes in performance, and determine performance satisfaction. The Turkish cultural adaptation, validity, and reliability of this measurement tool were carried out by Torpil, with an internal consistency coefficient ranging from 0.9 to 1.
Occupational Balance Questionnaire-11 (OBQ11-T) | From enrollment to the end of treatment at 4 weeks
  The task was used to evaluate occupational balance. The Occupational Balance Questionnaire is a questionnaire in which a person evaluates their occupational balance in relation to their current situation and daily life.
Stroke Impact Scale 3.0 | From enrollment to the end of treatment at 4 weeks
  The quality of life was evaluated with The Stroke Impact Scale. It is a self-report questionnaire that evaluates disability and health-related quality of life after stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri city hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.